CLINICAL TRIAL: NCT04472182
Title: Efficacy of Fluoride Varnish Containing Xylitol Coated Calcium Phosphate Versus Conventional Fluoride Varnish in Management of Hypersensitivity of Exposed Root Surfaces in Adult Patients: A Randomized Clinical Trial
Brief Title: Efficacy of Fluoride Varnish Containing Xylitol Coated Calcium Phosphate Versus Conventional Fluoride Varnish in Management of Hypersensitivity of Exposed Root Surfaces in Adult Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Peter Edward Ibrahim Abdelmalik, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoUniv
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Phosphates

STUDY DESIGN:
Intervention Model Description: Dentin Hypersensitivity
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride varnish with xylitol coated calcium and phosphate (Experimental)
  Interventions: Drug: Fluoride varnish with xylitol coated calcium and phosphate
- Conventional Fluoride varnish (Active Comparator)
  Interventions: Drug: Fluoride varnish with xylitol coated calcium and phosphate

INTERVENTIONS:
Drug: Fluoride varnish with xylitol coated calcium and phosphate — Fluoride varnish with xylitol coated calcium and phosphate

SUMMARY:
This clinical trial will be conducted to compare the efficacy of fluoride varnish containing xylitol coated calcium and phosphate or potassium nitrate gel versus conventional fluoride varnish in the management of hypersensitivity of non-carious exposed root surfaces in adult patients over a 12 months period.

ELIGIBILITY:
Inclusion Criteria of participants:

Males or females. Age: 20-50 years old. Patients having at least one tooth with exposed root surface Teeth with hypersensitivity, VAS ≥5 Patients with good oral hygiene. Co-operative patients who show interest to participate in the study

Exclusion criteria of participants:

Patients with bad oral hygiene Patients with orthodontic appliances, or bridge work that might interfere with evaluation Patients who are allergic to any ingredients will be used in the study. Carious teeth Mobile teeth. (Grade 2 or Grade 3) Teeth with hypersensitivity, VAS <5 Patients with physical disabilities Pregnant or lactating women Other dental defects that causes pain. Allergy from any used materials or any allergic reaction during our clinical trial (The trial will be stopped at once and all the needed management against any allergic reaction will be done.)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Pain due to Dentin Hypersensitivity | Two minutes before intervention
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale
Pain due to Dentin Hypersensitivity | 4 hours
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale
Pain due to Dentin Hypersensitivity | 2 days
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale
Pain due to Dentin Hypersensitivity | 4 months
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale
Pain due to Dentin Hypersensitivity | 8 months
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale
Pain due to Dentin Hypersensitivity | 12 months
  Pain arising from Dentin Hypersensitivity on exposed root surfaces using air blast measured by 10 cm VAS scale

SECONDARY OUTCOMES:
Measuring Salivary pH | Two minutes before intervention
  measuring Unstimulated Salivary pH using pH meter from 0-14
Measuring Salivary pH | 4 hours
  measuring Unstimulated Salivary pH using pH meter from 0-14
Measuring Salivary pH | 2 days
  measuring Unstimulated Salivary pH using pH meter from 0-14
Measuring Salivary pH | 4 months
  measuring Unstimulated Salivary pH using pH meter from 0-14
Measuring Salivary pH | 8 months
  measuring Unstimulated Salivary pH using pH meter from 0-14
Measuring Salivary pH | 12 months
  measuring Unstimulated Salivary pH using pH meter from 0-14
Image analysis to assess amount of plaque adherence | 2 minutes before intervention
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface
Image analysis to assess amount of plaque adherence | 4 hours
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface
Image analysis to assess amount of plaque adherence | 2 days
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface
Image analysis to assess amount of plaque adherence | 4 months
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface
Image analysis to assess amount of plaque adherence | 8 months
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface
Image analysis to assess amount of plaque adherence | 12 months
  Calculating the percentage (0%-100%) of area with plaque adherence in relation to the total area of the tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Abdelmalik, Master, Principal Investigator — Cairo University
Locations (1):
- Cairo U, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided